CLINICAL TRIAL: NCT04482855
Title: Low-level Laser in Treatment of Head and Neck Chronic Lymphedema: A Pilot Randomized Controlled Trial
Brief Title: Low-Level Laser in Head and Neck Chronic Lymphedema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Principal Investigator, Jie Deng, Associate Professor, PhD, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UPCC 01320
Record Dates: First submitted 2020-06-24; First posted 2020-07-23 (Actual); Results first posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-10

CONDITIONS: Head and Neck Cancer; Lymphedema; Fibrosis
MeSH Terms: conditions — Head and Neck Neoplasms; Lymphedema; Fibrosis | interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: Randomized, wait-list control
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Group 1 (laser group) (Experimental): Group 1 (laser group): After completion of the baseline measurements, Group 1 participants will be scheduled for LLLT. After completion of LLLT, participants will be scheduled for the 4-week and 8-week follow up data collection.
  Interventions: Device: Low-level laser
- Group 2 (wait-list control group) (No Intervention): Group 2 (wait-list control group): Group 2 participants will not undergo LLLT therapy but will complete all the same study assessments as the laser therapy group, including the baseline, and follow-up assessments. After the 8-week follow-up assessment, participants will be offered the same LLLT as the laser group.

INTERVENTIONS:
Device: Low-level laser — Low-level laser therapy
  Arms: Group 1 (laser group)

SUMMARY:
The purpose of this study is to evaluate the effect of low-level laser treatment (LLLT) on the severity of lymphedema, symptom burden, functional status, and quality of life in HNC survivors.

DETAILED DESCRIPTION:
Primary aim: To determine the impact of LLLT, as compared to wait-list control, on changes in severity of lymphedema.

Secondary aim: To determine the impact of LLLT, as compared to a wait-list control, on lymphedema-related symptom burden (e.g., tightness), functional impairments (e.g., range of motion in jaw and neck), and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* >6 months post HNC treatment
* No evidence of cancer confirmed with imaging tests
* Having head and neck lymphedema with or without fibrosis
* Completion of initial lymphedema therapy
* Lymphedema duration between 3-24 months
* Ability to speak and read English
* Ability to provide informed consent

Exclusion Criteria:

Patients will be excluded if they have any of the following medical conditions that would prohibit the safe implementation of LLLT:

* Pregnancy
* Acute infection
* Photosensitivity
* Chronic inflammatory diseases
* Venous thrombosis
* Carotid artery stenosis
* History of severe trauma
* Medication that affects body fluid and electrolyte balance
* Use of high doses of non-steroidal anti-inflammatory drugs
* Pre-existing skin rash, ulceration, open wound in the treatment area
* Active lymphedema therapy or physical therapy
* Allergic and other systemic skin diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-08-19 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania Abramson Cancer Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1 (Laser Group) | Group 2 (Wait-list Control Group)
Started | 12 | 13
Completed | 9 | 13
Not Completed | 3 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrew from the study before attending the study intervention sessions due to unexpected job duty | 1 | 0
Not completed — Withdrew from the study before attending the study intervention sessions due to new cancer diagnosis | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 (Laser Group) | Group 2 (Wait-list Control Group) | Total
Number analyzed (Participants) | 12 | 13 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.5 (5.06) | 62.3 (6.01) | 61.0 (5.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 10 | 12 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 12 | 12 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 13 | 25

OUTCOME MEASURES:

1. Primary Outcome: Total Severity of External Lymphedema and Fibrosis (LEF)
Description: Head and Neck Lymphedema and Fibrosis Assessment Criteria
  Change in total severity of external LEF from baseline to 8-week post-intervention visits. A larger change in this score means more reduction in the severity of external LEF.
  External LEF is measured by HN-LEF Assessment Criteria. The total external LEF severity score is calculated by summing the severity score of each site (total 9 sites, severity score ranging from 0-27). For each site, the severity of LEF includes no LEF (=0), mild (=1), moderate (=2), and severe (=3).
Time Frame: Baseline, 8-week post-intervention visit
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1 (Laser Group) | Group 2 (Wait-list Control Group)
Number analyzed (Participants) | 12 | 13
score on a scale
  Total severity score of LEF at baseline visit | 5.42 (2.07) | 4.08 (2.33)
  Total severity score of LEF at 8-week post-intervention visit | 3.22 (1.86) | 4.62 (1.71)

2. Secondary Outcome: Symptom Burden Score: Soft Tissues and Neurologic Toxicity Subscale
Description: Head and Neck Lymphedema and Fibrosis Symptom Inventory
  Change in symptom burden score from baseline to 8-week post-intervention. A larger change in this score means decreased symptom burden.
  Symptom burden is assessed by Head and Neck Lymphedema and Fibrosis Symptom Inventory (HN-LEF SI). Higher scores (score ranging from 0-5) indicate increased symptom burden. There are 7 subscales and only one subscale (Soft Tissues and Neurologic Toxicity) score is reported here.
Time Frame: Baseline, 8-week post-intervention visit
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1 (Laser Group) | Group 2 (Wait-list Control Group)
Number analyzed (Participants) | 12 | 13
score on a scale
  Soft Tissues and Neurologic Toxicity at baseline | 2.46 (0.97) | 1.63 (1.03)
  Soft Tissues and Neurologic Toxicity at 8-week post-intervention visit | 1.73 (1.32) | 1.23 (0.92)

3. Secondary Outcome: Neck Range of Motion Degree: Right Lateral Rotation
Description: Change in neck range of motion degree from baseline to 8-week post-intervention. A larger change in this degree means better outcome with increased neck range of motion.
  Cervical Range of Motion Device, a valid and reliable tool, was used to measure the amount of neck movement (degrees) for the following neck movements: forward flexion, extension, right and left lateral flexion, and right and left rotation. Only right lateral rotation is reported here.
Time Frame: Baseline, 8-week post-intervention visit
Measure: Mean (Standard Deviation); unit: degrees of neck movements
Arm/Group | Group 1 (Laser Group) | Group 2 (Wait-list Control Group)
Number analyzed (Participants) | 12 | 13
degrees of neck movements
  Right lateral rotation at baseline visit | 45.38 (13.54) | 48.04 (6.98)
  Right lateral rotation at 8-week post-intervention visit | 52.78 (11.18) | 47.85 (10.92)

4. Secondary Outcome: Quality of Life Score: Feeding Tube
Description: EORTC QLQ-H&N35 was used to assess HNC-related quality of life.
  Change in EORTC QLQ-H&N35 score from baseline to 8-week post-intervention. A larger reduction in this score means decreased symptom burden and better quality of life.
  The HNC-specific EORTC QLQ-H&N35 module is a supplement, containing seven multi-item scales (pain, swallowing, senses problems, speech problems, trouble with social eating and social contact, and less sexuality) and eleven single-item scales (teeth, opening mouth, dry mouth, sticky saliva, coughing, felt ill, pain killers, nutritional supplements, feeding tube, weight loss, weight gain). The QLQ-H&N35 scale employs a 4-point response format (''not at all" to ''very much"). Scale scores are transformed to a scale from 0 to 100 according to the EORTC scoring algorithm. For the symptoms scales, a higher score indicates a higher level of symptom burden. Only feeding tube scale is reported here.
Time Frame: Baseline, 8-week post-intervention visit
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1 (Laser Group) | Group 2 (Wait-list Control Group)
Number analyzed (Participants) | 12 | 13
score on a scale
  Quality of life -feeding tube scale score at baseline visit | 16.67 (38.92) | 15.38 (37.55)
  Quality of life -feeding tube scale score at 8-week post-intervention visit | 0 (0) | 7.69 (27.74)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the baseline visit to 8-week post-intervention visit.
Description: Common Terminology Criteria for Advance Events (CTCAE) version 5.0 was used to evaluate adverse events of the trial.
Arm/Group | Group 1 (Laser Group) | Group 2 (Wait-list Control Group)
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/13
Other Adverse Events (participants affected / at risk) | 0/12 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-12): https://cdn.clinicaltrials.gov/large-docs/55/NCT04482855/Prot_SAP_000.pdf